CLINICAL TRIAL: NCT03767257
Title: A Phase 2 Study of Colesevelam for Lenalidomide-Associated Diarrhea
Brief Title: A Study of Colesevelam for Lenalidomide-Associated Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-421
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma; Diarrhea
Keywords: Lenalidomide Associated Diarrhea; Colesevelam; 18-421; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Multiple Myeloma; Diarrhea | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Myeloma (Experimental): Individuals with Myeloma on lenalidomide maintenance who experience grade 2 or more diarrhea
  Interventions: Drug: Colesevelam Pill

INTERVENTIONS:
Drug: Colesevelam Pill — For treatment with colesevelam, the starting dose will be 1250 mg (2 x 625 mg) with food which can be increased to 6 tablets max per day based on efficacy and tolerability. Coleveselam should not be taken within 4 hours before or after lenalidomide and other interacting medications. All participants will be given a pill diary to record intake of colesevelam. The effect of colesevelam on lenalidomide-associated diarrhea will be evaluated after 1, 2, 4, 12 weeks after start of treatment. If the diarrhea does not respond to the starting dose of colesevelam, the dose can be increased every 2 days to 2 tablets two times per day (2 x 625 mg BID) and later to 3 tablets two times per day (3 x 625 mg BID). The colesevelam dose can be decrease to 1 tablet per day if there has been improvement of diarrhea but emergence of side effects.

SUMMARY:
The purpose of this study is to test the safety of colesevelam and find out what effects, if any, colesevelam has on lenalidomide associated diarrhea in participants with multiple myeloma on lenalidomide maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Memorial Sloan Kettering Cancer Center (MSK) confirmed diagnosis of multiple myeloma
* Treatment with single agent lenalidomide maintenance
* Patient must be >/= 18 years of age at the time of informed consent
* Experiencing grade 1 or more diarrhea according to the CTCAE 5.0 criteria for at least 4 out of 7 days preceding screening and study inclusion
* Scheduled to receive lenalidomide maintenance cyles at MSK
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Patients with history of bowel obstruction
* Patients with serum triglyceride levels >300 mg/dL
* Patients wit history of hypertriglyceridemia-induced panreatitis
* Patients with known hypersensitivity to colesevelam or any component to the formulation
* Patients currently already receiving a bile acid sequestrant or have previously used bile acid sequestrant drugs for diarrhea and had no benefit
* Patients with diarrhea secondary to infection. Stool studies for GI pathogens should be collected prior to starting colesevelam but do not need to be resulted prior to starting Day 1 dose of colesevelam, unless infection is suspected by the treating investigator, in which case (Clostridium difficile PCR when clinically indicated, GI pathogen panel, stool ova and parasites, Giardia and Cryptosporum stool antigen tests will need to be resulted at investigator discretion.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malin Hultcrantz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Myeloma
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Myeloma
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 60 [47 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement of Lenalidomide-associated Diarrhea Evaluated by CTCAE 5.0
Description: To evaluate the ability of colesevelam to improve lenalidomide-associated diarrhea in participants with multiple myeloma treated with lenalidomide maintenance. Diarrhea will be evaluated using Common Terminology Criteria for Adverse Events (CTCAE) grading. The primary end-point is improvement of diarrhea to grade 1 or better according to the CTCAE 5.0 scale by 4 weeks of treatment with colesevelam.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Myeloma
Number analyzed (Participants) | 25
Participants
  Improvement by at least 1 grade per CTCAE scale | 22
  Did not respond to colesevelam treatment | 3

2. Secondary Outcome: Number of Participants With GI Symptom Assessment
Description: To assess GI symptoms using Patient Reported Outcomes within the Common Terminology Criteria for Adverse Events
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Myeloma
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Participants With Myeloma
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 25/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Myeloma (N=25)
Diarrhea (Gastrointestinal disorders) | 25
Constipation (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Acid reflux (Gastrointestinal disorders) | 1
Shingles (Infections and infestations) | 1
Sars-CoV-2 (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT03767257/Prot_SAP_000.pdf